CLINICAL TRIAL: NCT02211456
Title: Dual Site Left Endocardial Pacing for Cardiac Resynchronisation Therapy
Brief Title: An Assessment of Dual Site Left Ventricular Endocardial Pacing
Acronym: DOUBLE-CRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Dr James Gamble, Research Fellow, Oxford University Hospitals NHS Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DOUBLE-CRT_72014
Record Dates: First submitted 2014-08-01; First posted 2014-08-07 (Estimated); Results first posted 2021-03-04 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-02

CONDITIONS: Atrial Fibrillation; Ventricular Tachycardia; Heart Failure
Keywords: Endocardial pacing; Multi site pacing
MeSH Terms: conditions — Atrial Fibrillation; Tachycardia, Ventricular; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Participants (Experimental): Having an ablation procedure with access to the left side of the heart
  Interventions: Procedure: Atrial Fibrillation/flutter (AF) or Ventricular Tachycardia (VT) ablation with multi-site pacing protocol

INTERVENTIONS:
Procedure: Atrial Fibrillation/flutter (AF) or Ventricular Tachycardia (VT) ablation with multi-site pacing protocol — Pacing at several endocardial sites in isolation and individually will be performed, with response to this assessed by LV dp/dt max

SUMMARY:
We are investigating ways to help patients with heart failure, which is caused by damaged hearts which function less well, and cause symptoms of breathlessness, fatigue, lack of energy and swelling.

Cardiac Resynchronisation Therapy (CRT) pacemakers are used to improve the pumping function of the main heart chamber in certain suitable people with heart failure. CRT requires a pacemaker with 2 wires, one placed inside the right heart chamber and one normally placed on the outside of the left heart chamber. These two wires act together to re-time the coordination of the heartbeat, which is known to improve heart function.

The investigators are assessing whether they might be able to improve heart function even more by placing two wires on the inside of the left heart chamber, rather than one around the outside.

The investigators wish to assess whether:

1. Using two wires within the left side of the heart gives a greater increase in heart function than one.
2. It is possible to choose the best spot inside of the heart by measuring the pattern of the heart beat.
3. Is it possible to use a different type of heart monitor placed outside the body instead of a monitor wire inside the heart to assess improvement in heart function? They are investigating this in people with hearts that beat less effectively than normal.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 60 years or above.
* Having a suitable Atrial Fibrillation/flutter or Ventricular Tachycardia ablation procedure
* Evidence of abnormal Left Ventricular structure and function, as shown by Left Ventricular ejection fraction of less than 40%

Exclusion Criteria:

* Severe peripheral vascular disease (that would make arterial access more risky)
* Haemodynamic instability (such that a longer procedure is inadvisable)

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-12; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim R Betts, MD, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (1):
- Oxford University Hospitals NHS Trust, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Background] Bordachar P, Derval N, Ploux S, Garrigue S, Ritter P, Haissaguerre M, Jais P. Left ventricular endocardial stimulation for severe heart failure. J Am Coll Cardiol. 2010 Aug 31;56(10):747-53. doi: 10.1016/j.jacc.2010.04.038. PMID 20797486
- [Background] Shetty AK, Sohal M, Chen Z, Ginks MR, Bostock J, Amraoui S, Ryu K, Rosenberg SP, Niederer SA, Gill J, Carr-White G, Razavi R, Rinaldi CA. A comparison of left ventricular endocardial, multisite, and multipolar epicardial cardiac resynchronization: an acute haemodynamic and electroanatomical study. Europace. 2014 Jun;16(6):873-9. doi: 10.1093/europace/eut420. Epub 2014 Feb 12. PMID 24525553
- [Background] Rogers DP, Lambiase PD, Lowe MD, Chow AW. A randomized double-blind crossover trial of triventricular versus biventricular pacing in heart failure. Eur J Heart Fail. 2012 May;14(5):495-505. doi: 10.1093/eurjhf/hfs004. Epub 2012 Feb 6. PMID 22312038
- [Background] Betts TR, Gamble JH, Khiani R, Bashir Y, Rajappan K. Development of a technique for left ventricular endocardial pacing via puncture of the interventricular septum. Circ Arrhythm Electrophysiol. 2014 Feb;7(1):17-22. doi: 10.1161/CIRCEP.113.001110. Epub 2014 Jan 14. PMID 24425419

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants: Having an ablation procedure with access to the left side of the heart
  Atrial Fibrillation/flutter (AF) or Ventricular Tachycardia (VT) ablation with multi-site pacing protocol: Pacing at several endocardial sites in isolation and individually will be performed, with response to this assessed by LV dp/dt max
  All patients underwent the pacing protocol
Period: Overall Study
Arm/Group | Participants
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Participants
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15
Region of Enrollment [Number; unit: participants]
  United Kingdom | 15
Ischaemic aetiology of left ventricular dysfunction [Count of Participants; unit: Participants] | 12
Left ventricular ejection fraction [Mean (Standard Deviation); unit: %] | 27 (8)

OUTCOME MEASURES:

1. Primary Outcome: Acute Haemodynamic Response to Dual Left Ventricular Pacing
Description: Acute haemodynamic response to pacing (change in Left Ventricular dP/dt max) between dual site Left Ventricular pacing and biventricular pacing Pacing protocols were performed with a baseline of 30 seconds of right ventricular pacing followed by two 30-second test configurations, and then a further baseline. The pacing configurations were tested, in a randomized order, 3 times each.
  Electrophysiology catheters were positioned at the right ventricular mid septum for baseline pacing, and at the left ventricular septum and at the left ventricular lateral wall, at the site of latest electrical activation i identified from a left ventricular electrical activation map This provided two single-site left ventricular pacing configurations, which could be combined to allow right ventricular and left ventricular lateral (Biventricular pacing) and left ventricular septal and left ventricular lateral (dual left ventricular pacing)
Time Frame: Mean of multiple recordings in each patient as detailed above
Measure: Mean (95% Confidence Interval); unit: % difference
Arm/Group | Participants
Number analyzed (Participants) | 15
% difference | 3.7 [1.0 to 6.3]
Statistical Analysis 1: Comparison: Participants; The data derived from this study was complex multi-level data with errors due to patient-level and intra-patient repeat factors. Accordingly, we used generalized multi-level modelling (GLMM) with random effects; Test type: Superiority; p < 0.05, Mixed Models Analysis; Mean Difference (Final Values) = 3.7, 95% CI 2-sided [1 to 6.3]

ADVERSE EVENTS:
Arm/Group | Participants
Serious Adverse Events (participants affected / at risk) | 1/15
Other Adverse Events (participants affected / at risk) | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants (N=15)
Stroke (Nervous system disorders) | 1 (1) — One patient developed neurological symptoms shortly after waking up from anesthesia after his ventricular tachycardia ablation and was found to have had a left sided stroke.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes